CLINICAL TRIAL: NCT05705648
Title: Nutritional Management of Post COVID-19 Cognitive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00109795
Record Dates: First submitted 2023-01-27; First posted 2023-01-31 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Long COVID
Keywords: brain fog; confusion; memory loss; functional decline
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue; Confusion; Memory Disorders | interventions — Safflower Oil

STUDY DESIGN:
Intervention Model Description: Randomised placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Medium chain triglyceride oil 15ml tid x 5 months
  Interventions: Dietary Supplement: medium chain triglyceride oil
- Placebo (Placebo Comparator): Safflower oil 15mls tid x 5 months
  Interventions: Dietary Supplement: Safflower oil

INTERVENTIONS:
Dietary Supplement: medium chain triglyceride oil — Medium chain triglyceride oil
  Arms: Intervention
Dietary Supplement: Safflower oil — Safflower oil
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about in brain "fog" complaints associated with long-COVID in people aged 22-50-years. The main questions it aims to answer are:

* the natural course of brain "fog" complaints
* the effect, if any of supplemental dietary oil on brain "fog" complaints Participants will be asked to undergo some brain testing (X-rays and questions. Treatments they'll be given will be one of two supplemental oils to consume daily.

Researchers will compare outcomes in the two different oil groups to see if it has any effect on brain "fog" complaints.

DETAILED DESCRIPTION:
Randomized placebo-control clinical trial comparing two types of nutritional oil and evaluating the impact, if any, on subjective complaints of long-COVID cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

* confirmed COVID infection, at least 3 months previously, with ongoing cognitive complaints
* all other medical conditions stable, and on stable doses of medications (if required)

Exclusion Criteria:

* COVID infection not confirmed by PCR or Rapid test
* unable to speak English
* pre-COVID cognitve complaints, and/or medical diagnoses affecting cognitive function

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Cognigram(R) | 12-months
  computer-based cognitive test

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | 12-months
  Cognitive test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No